CLINICAL TRIAL: NCT04267861
Title: Retrospective Study of M7824 Related Adverse Effects in Adults With Cancer
Brief Title: M7824 Related Adverse Effects in Adults With Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999920055; 20-C-N055
Record Dates: First submitted 2020-02-12; First posted 2020-02-13 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-04-16

CONDITIONS: Neoplasms; Skin Neoplasms
Keywords: Skin Neoplasms; Immunotherapy; Anti-PD-1; Natural History
MeSH Terms: conditions — Neoplasms; Skin Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Medical records of subjects enrolled on NCI protocols 15-C-0179 and 18-C-0056

SUMMARY:
Background:

Immunotherapy drugs use a person s own immune system to help fight cancer. These drugs work better for some people than others. The drug M7824 has helped some people with cancer. But it can cause side effects. Researchers want to learn all the side effects that M7824 can cause. Once they do, they can prevent or reduce these side effects in future cancer treatments. This will lead to better overall outcomes for people with cancer.

Objective:

To make a thorough list of adverse events in people with cancer being treated with systemic therapies including M7824 at the National Cancer Institute (NCI).

Eligibility:

Participants previously enrolled in NCI protocols #15-C-0179 and #18-C-0056

Design:

All needed data have already been collected. These data are stored in existing records and databases.

Researchers will review the medical records of adults with cancer who were enrolled in the above protocols. The data collected will be relevant to the specific objectives being addressed.

Data will be collected only if 2 conditions are met. One, the principal investigator gave permission for use of the data gathered in the trial. Two, the participants of the trial did not opt out of future use of the data.

Other protocols may be added. This will be done with an amendment.

...

DETAILED DESCRIPTION:
Immunotherapy agents utilize the immune system to help fight cancer. A number of immunotherapy drugs have been approved for use in certain cancers. Despite being effective in some patients, many of these promising drugs do not demonstrate efficacy in other patients. M7824 (MSB0011359C), a bifunctional fusion protein that blocks both PD-L1 and transforming growth factor beta (TGF-beta) signaling, is a promising novel drug that has proven efficacious in a subset of cancer patients. However, we have observed side effects in patients receiving M7824 that include both immune related adverse events and skin neoplasms. It is imperative that these M7824 side effects be identified and characterized so that they can be prevented or diminished during future cancer treatments. By thoroughly analyzing the side effect profile of this drug, management of adverse effects and overall patient outcomes can be better understood and optimized.

The primary goal of this protocol is to perform a retrospective chart review for the investigation of the adverse events arising in cancer patients being treated with systemic therapies including M7824 at the National Cancer Institute (NCI). This study will not involve the use of specimens or participant contact. All data that are needed have already been collected on the individual treatment protocols and are available in CRIS records or protocol specific databases. Data will only be collected from treatment protocols where the PI has given permission for use of the data on the trial the subjects were enrolled on and the subjects did not opt out of future use of data. This protocol will be amended to incorporate new research objectives and new protocols as necessary.

ELIGIBILITY:
* INCLUSION CRITERIA:

Adults with cancer enrolled on immunotherapy treatment protocols including M8724 in the NCI.

EXCLUSION CRITERIA:

Patients who opted out of future use of data on their prior studies will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects enrolled on CC protocols 15-C-0179 and 18-C-0056
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
M7824 related adverse events | ongoing
  adverse event frequency and characterization

CONTACTS AND LOCATIONS:
Overall Officials: Isaac F Brownell, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States